CLINICAL TRIAL: NCT05159258
Title: Morphological Analysis and Classification of Posterior Malleolar Fractures Based on CT Scans
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Hailin Xu, Associate Professor, Peking University People's Hospital
Other Study IDs: MACPMFCTscans
Record Dates: First submitted 2021-11-18; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Morphological Analysis and Classification; Posterior Malleolar Fractures; CT Scans
Keywords: Ankle fractures; Posterior malleolar fractures; Classification; Mechanism
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:

SUMMARY:
The study was to propose a classification system of posterior malleolar fractures by fracture lines with the use of CT scans, including 3D CT reconstruction, which can better understand morphological characteristics, analyze the mechanism and guide the surgeon to choose optimal approach and fixation.

DETAILED DESCRIPTION:
The investigators retrospectively analyzed consecutive patients with ankle fractures from January 2013 and December 2019 . Participants were included with OTA/AO type 44 fractures involving posterior malleolus and CT scans. The exclusion criteria were: (1) previous ankle surgery; (2) pathological fractures; (3) previous deformity in ankle joint; (4) age ≤16 years old. Finally, A total of 128 patients were included in this study. 128 consecutive participants with posterior malleolar fractures from January 2013 and December 2019. CT data were loaded into Mimics software (V20.0, Materialize), in which 3D CT reconstruction, morphological analysis and data measurements were made. Statistical analysis was performed using the Statistical Packages for Social Sciences V23.0 (SPSS, Chicago, IL, USA). Mann-Whitney U test were used. P value of < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* OTA/AO type 44 fractures involving posterior malleolus and CT scans

Exclusion Criteria:

* Previous ankle surgery
* Pathological fractures
* Previous deformity in ankle joint
* Age ≤16 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: OTA/AO type 44 fractures involving posterior malleolus
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
posterior malleolar fracture classification | 2013-2019
  Haraguchi, Bartonicek and Mason & Molloy classification
area of posterior malleolar fragment | 2013-2019
area of remaining stable plafond | 2013-2019
length of remaining fibular notch | 2013-2019
length of involving fibular notch | 2013-2019

IPD SHARING:
Plan to Share IPD: Yes
The results of the study are publicly available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code